CLINICAL TRIAL: NCT05972915
Title: Separation Sign: New Ultrasound Sign to Rule Out Diagnosis of Placenta Accreta
Brief Title: Separation Sign: New Ultrasound Sign to Rule Out Placenta Accreta
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Other Study IDs: Separation sign
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Accreta, Placenta
Keywords: placenta accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Separation sign — The separation sign was recorded as positive if separation of the myometrium from the placenta was observed in all areas of the placenta. The sign was recorded as negative if the myometrium and placenta moved as one structure and no clear zone could be seen over any part of the placenta after release, even if separation was noted at the margins of the placenta.

SUMMARY:
To assess the 'separation sign' as a predictor of normal placental separation in a large cohort of women at risk for placenta accrete spectrum and in a high-risk subgroup with placenta previa or anterior low-lying placenta and have history of at least one previous Cesarean delivery.

DETAILED DESCRIPTION:
A prospective Observational Cohort study The study population includes high-risk cohort of women was defined as those who had placenta previa or an anterior low-lying placenta, in addition to at least one previous Cesarean delivery. They will be asked to participate in the study after been evaluated to ensure fulfilling inclusion and exclusion criteria.

Women will be enrolled in the study after giving written informed consent

The patients will be submitted to:

**Full history taking including: Details of gestational age at the time of scanning, maternal age and risk factors , history of dilatation and curettage, in-vitro fertilization and other previous uterine surgery were assessed.

***Detailed trans-abdominal sonographic examination of the placenta was performed, assessing standard ultrasound markers of PAS. Two experienced sonographic operators performed all examinations using (Toshiba Xario 200) with 3D/4D curved-array trans-abdominal transducer (4-8.5 MHz). All examinations were performed with a full bladder, defined as a volume between 250mL 500mL quantified using the inbuilt ellipsoid volume calculation.

To assess for the separation sign, pressure was applied using an ultrasound probe so that the hypoechoic retroplacental clear zone normally observed between the placenta and myometrium disappeared. The pressure was then rapidly released in order to generate the force required to see movement. On release, in cases with normal placentation, the non-elastic placenta keeps moving away from the probe after the highly elastic myometrium has 'snapped' back into place. This sometimes causes the placenta either to keep moving briefly or even to 'bounce' and leads to the appearance or enhancement of the clear zone. With a negative separation sign, no separate movement of the placenta from the myometrium can be seen. The separation sign was recorded as positive if separation of the myometrium from the placenta was observed in all areas of the placenta. The sign was recorded as negative if the myometrium and placenta moved as one structure and no clear zone could be seen over any part of the placenta after release, even if separation was noted at the margins of the placenta. Classification into positive or negative separation sign was highly stringent and, in case of any doubt, the result was recorded as uncertain. The latter occurred most often when the images obtained were suboptimal, for example, owing to tissue attenuation, high body mass index (BMI) or significant scarring. If women were scanned on multiple occasions, the separation sign result obtained closest to 28 weeks' gestation was used in order to minimize differences in scanning over the course of gestation.

***Based on histopathology results in cases in which hysterectomy was performed. A diagnosis of PAS was excluded if the placenta separated spontaneously at delivery, was delivered by controlled cord traction or was delivered by simple manual removal. Histopathological analysis was carried out by a pathologist with expertise in PAS, with the specific sampling site marked by the surgical team according to intrapartum findings. The pathologists were blinded to the separation sign classification but not to surgical findings.

ELIGIBILITY:
Inclusion Criteria:

* History of previous cesarean section or hysterotomy.

  * Placenta previa or low lying anterior placenta.
  * From 28 wks to Full term.

Exclusion Criteria:

1. Multiple pregnancies.
2. Medical disorder as diabetes mellitus, hypertension. 3. Obese patients. BMI > 30 4. Intrauterine growth retardation.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The study population includes high-risk cohort of women was defined as those who had placenta previa or an anterior low-lying placenta, in addition to at least one previous Cesarean delivery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
separation sign | 1 month before delivery
  The separation sign was recorded as positive if separation of the myometrium from the placenta was observed in all areas of the placenta. The sign was recorded as negative if the myometrium and placenta moved as one structure and no clear zone could be seen over any part of the placenta after release, even if separation was noted at the margins of the placenta.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided